CLINICAL TRIAL: NCT01515267
Title: Automated Left Ventricular Function Evaluation by LVivoEF
Acronym: LVivoEF
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: DiA Imaging Analysis Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: DIA100
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: EF Evaluation From 4 Chamber Plane; EF Evaluation From 2 Chamber Plane; Biplane EF Evaluation; Left Ventricular Function
Keywords: EF; EDV; ESV; Biplane; Echocardiography

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Left ventricular ejection fraction (EF) is evaluated in every echocardiographic examination either by visual estimation (eyeballing) requiring high level of training and expertise and/or by manual tracing of the endocard from which EF is calculated (manual biplane method (MBP)). This procedure is subjective and time consuming. The objective of this study is to compare the performance of LVivoEF software system to the measurements obtained by the routinely used methods.

DETAILED DESCRIPTION:
LVivoEF is a decision support system (software) for automated global left ventricle (LV) systolic function evaluation from echocardiographic examinations. LVivoEF technology is based on a novel image processing algorithm for LV edge detection and ejection fraction (EF) evaluation. LVivoEF provides fully automated measurements of the left ventricle (LV) from two apical views the four chamber (4CH) and the two chamber (2CH).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Patients referred to an echocardiographic examination. The patients will be consecutive until 30% of patients with normal LV function are enrolled. After that only consecutive patients with abnormal LV function will be included.

Exclusion Criteria:

* Examinations in which more than one third of the endocard is not visible in a plane (2CH/4CH)
* Patients with Left bundle branch block (LBBB)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients referred to an echocardiographic examination
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-11

CONTACTS AND LOCATIONS:
Overall Officials: Noah Liel-Cohen, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka university medical center, Beersheba, Israel